CLINICAL TRIAL: NCT03371576
Title: Comparison of Two Toric IOL´s With Different Haptic Design: Optical Quality After 1 Year
Brief Title: Clinical Analysis of Two Toric Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Michael Lasta, Principal investigator, Hospital Hietzing
Other Study IDs: HHietzing
Record Dates: First submitted 2017-11-23; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Cataract; IOL
Keywords: toric IOL
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2 different torical intraocular lenses
  Interventions: Device: intraocular lenses

INTERVENTIONS:
Device: intraocular lenses

SUMMARY:
Purpose: Comparison of two torical intraocular lenses with differents haptic design in patients with cataract.

Methods: In this prospective, randomized clinical trial 120 eyes of 60 patients underwent phacoemulsification. In patient's eyes the Tecnis torical IOL (Abbott Medical Optics) or the AT Torbi torical 709 MB IOL (Zeiss Medical AG) were randomly implanted. Three months after surgery visual acuity, rotation stability and astigmatism correction were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age related cataract on both eyes
* Corneal astigmatism 1,0- 4,0 D
* Potential postoperative visus 1,0
* No other ocular pathology as cataract
* Age 18 - 80
* Written informed consent to surgery and participation in the study

Exclusion Criteria:

* Pregnancy, breastfeeding
* Amblyopy, diabetic retinopathy, uveitis or other relevant ophthalmologic diseases
* Optical media disturbances due to: corneal and vitreal opacity, PEX
* Irregular astigmatism measured with corneal topography (Visante-omni), keratoconus
* ≥ 10 degrees difference between the axis of keratometry measurement of the IOL Master and the simulated K reading of the corneal topograph (Visante-omni)
* Trauma, ocular surgery performed within 6 months
* Traumatic cataract
* Potential postoperative visus under 1,0

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cataract on both eyes.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
uncorrected visual acuity | 1 year
  visual acuity in logMARon an ETDRS Chart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mihaltz K, Lasta M, Burgmuller M, Vecsei-Marlovits PV, Weingessel B. Comparison of Two Toric IOLs with Different Haptic Design: Optical Quality after 1 Year. J Ophthalmol. 2018 Feb 11;2018:4064369. doi: 10.1155/2018/4064369. eCollection 2018. PMID 29607216